CLINICAL TRIAL: NCT00704600
Title: A Phase I/II Trial Testing Nelfinavir, an Inhibitor of Akt Signaling, in Combination With Preoperative Chemoradiotherapy in Patients With Locally Advanced Rectal Cancer
Brief Title: Nelfinavir, a Phase I/Phase II Rectal Cancer Study
Acronym: Nelfinavir
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEC 07-03-026
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Colorectal Cancer; Colorectal Carcinoma; Colorectal Tumors; Neoplasms, Colorectal
Keywords: Locally advanced rectal cancer; nelfinavir; radiosensitivity; chemoradiation
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Nelfinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- nelfinavir (Experimental): see intervention
  Interventions: Drug: nelfinavir

INTERVENTIONS:
Drug: nelfinavir — Phase I:
  * take nelfinavir tablets (minimum 6, maximum 10) starting 7 days before start of chemoradiotherapy, for 45 days
  * day 0 and day 7 and week 2-3-4-5-6-7 weekly blood sample
  * day 0: PET-CT
  Phase II:
  * take nelfinavir tablets (MTD from phase 1) starting 7 days before start of chemoradiotherapy, for 45 days
  * day 0 and day 7 and week 2-3-4-5-6-7 weekly blood sample
  * day 7 biopsy
  * day 7, 21 and week 15 :PET-CT + perfusion CT
  Other Names: Viracept

SUMMARY:
The aim is to study safety and activity of nelfinavir , added to standard chemoradiotherapy in patients with locally advanced rectal cancer. Furthermore analysis of the effect of nelfinavir combined with chemoradiation on tumour tissue will be studied

DETAILED DESCRIPTION:
Objective of the study:

The aim is to study safety and activity of nelfinavir, added to standard chemoradiotherapy (28x1.8 Gy and capecitabine 825 mg/m2 BID) in patients with locally advanced rectal cancer. Furthermore analysis of the effect of nelfinavir combined with chemoradiation on tumor tissue will be studied.

Study design:

This is an open label, single-center phase I/II trial. During phase I the toxicity of 2 dose levels will be studied (750 mg BID and 1250 mg BID). During phase II the activity of nelfinavir in combination with capecitabine and radiotherapy will be studied, using the MTD from phase I. With respect to translational research, phosphorylation of Akt in monocytes and tumorcells will be measured at different timepoints during treatment. Furthermore, dynamic CT-PET scans will be obtained at different time points to get an impression of changes in SUV and perfusion during treatment and to correlate these changes with pathological response.

Study population:

Patients with locally advanced rectal cancer, who are candidates for chemoradiotherapy. In phase I, 6 patients will be included. In case of the occurrence of dose limiting toxicity, extra patients will be included, according to the rules described in the protocol. In phase II, 55 patients will be included.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the rectum (tumor <15cm from anal verge)
* Age >= 18 years
* UICC T3-4 N0-2 M0
* WHO performance status 0-2
* Less than 10 % weight loss the last 6 months
* No recent (< 3 months) severe cardiac disease (arrhythmia, congestive heart failure, infarction)
* Serum bilirubin = or < 3x normal
* ASAT and ALAT = or < 2,5x normal
* Creatinin clearance >50 ml/min
* Willing and able to comply with the study prescriptions
* No history of prior pelvic radiotherapy
* No known HIV infection
* No hemophilia
* No concurrent medication that is metabolized by the CYP3A4 isoenzyme (calcium channel blockers, antifungal agents, macrolide antibiotics, gastrointestinal prokinetics, terfenadin, midazolam)
* Statins should be stopped (except pravastatin and fluvastatin),
* No concurrent use of St. John's Wort (Hypericum perforatum)
* Women should not be pregnant or lactating
* Being willing and able to undergo one extra biopsy
* Have given written informed consent before patient registration

Exclusion Criteria:

* the opposite of the above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-09; Primary Completion 2010-09 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
phase I: Incidence of any grade 3 or higher non-hematological or grade 4 or higher hematological toxicity (CTCAE v3.0) and of grade 4 or higher postoperative toxicity within 30 days post-surgery phase II:rate of pathological complete remission | 22 wks

CONTACTS AND LOCATIONS:
Overall Officials: Ph. Lambin, MD PhD, Principal Investigator — Maastro Clinic, The Netherlands
Locations (1):
- Maastro clinic, Maastricht, Netherlands